CLINICAL TRIAL: NCT07100600
Title: An Open-label, Randomized, Controlled Trial of Trastuzumab Rezetecan Combined With Radiotherapy Versus Trastuzumab Rezetecan in the Treatment of HER2-positive Advanced Breast Cancer With Brain Metastases
Brief Title: Trastuzumab Rezetecan Combined With Radiotherapy Versus Trastuzumab Rezetecan in the Treatment of HER2-positive Advanced Breast Cancer With Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-408-001
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Advanced Breast Cancer; Brain Metastases; Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Trastuzumab Rezetecan
  Interventions: Drug: Trastuzumab Rezetecan
- experimental group (Experimental): Trastuzumab Rezetecan combined with radiotherapy
  Interventions: Drug: Trastuzumab Rezetecan; Radiation: FSRT or WBRT

INTERVENTIONS:
Drug: Trastuzumab Rezetecan — Trastuzumab Rezetecan：4.8mg/kg Q3W
Radiation: FSRT or WBRT — FSRT （8Gy/3-5 fx）or WBRT（30Gy/10fx）
  Arms: experimental group

SUMMARY:
A total of 224 subjects of HER2-positive advanced breast cancer with brain metastases are planned to be enrolled. Eligible subjects will be randomly assigned in a 1:1 ratio to the group receiving Trastuzumab Rezetecan combined with radiotherapy or the group receiving Trastuzumab Rezetecan monotherapy until disease progression, intolerable toxicity, withdrawal of informed consent, or the study determines that treatment must be terminated (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 yrs old;
2. Pathologically confirmed HER2-positive advanced breast cancer;
3. At least one measurable intracranial lesion according to RANO-BM criteria, which had not received local treatment;
4. Without prior cranial radiation and had no indication for immediate local treatment or refuse to local treatment;
5. Life expectancy is not less than 6 months.
6. Adequate function of major organs.

Exclusion Criteria:

1. Subjects with leptomeningeal metastasis
2. CNS complications requiring emergency neurosurgical intervention
3. Previous treatment with trastuzumab deruxtecan (DS-8201a) or any other antibody drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase 1 inhibitor;
4. Suffering from heart disease that is not well controlled or having clinical symptoms
5. History of clinically significant lung disease；
6. Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.
7. Female subjects during pregnancy and lactation
8. Any other conditions that researchers believe that patients are unsuitable for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 224 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2030-07-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 1.5 years

SECONDARY OUTCOMES:
CNS-ORR | 2 months
ORR by investigator using RECIST Guideline | 2 months
CNS-PFS | 1.5 year
Adverse events | up to 1.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Professor, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No